CLINICAL TRIAL: NCT06566755
Title: Study of Cadonilimab(AK104) Combined With Chemotherapy and Bevacizumab as First-line Treatment for RAS Mutated or Right Sided-metastatic MSS Colorectal Cancer
Brief Title: Cadonilimab (AK104) Combined With Chemotherapy and Bevacizumab as First-line Treatment for RAS Mutated or Right Sided-metastatic MSS Colorectal Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Caigang Liu (Other)
Responsible Party: Sponsor-Investigator, Caigang Liu, professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AK104-IIT-C-M-0020
Record Dates: First submitted 2024-08-21; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cadonilimab (AK104) combined with chemotherapy and bevacizumab (Experimental): Participants receive Cadonilimab PLUS chemotherapy and bevacizumab of each 21-day cycle.
  Treatment period (4-8 cycles)：
  * Cadonilimab: 10mg/kg, intravenous infusion, D1, Q3W;
  * CapeOx chemotherapy regimen Q3W+ bevacizumab, Q3W:
  oxaliplatin: 130 mg/m2 intravenous infusion, D1, Q3W capecitabine: 850 mg/m2 orally, D1-14, Q3W, twice daily; bevacizumab injection: 7.5mg/kg, IV, D1, Q3W. Maintenance treatment period：
  * Cadonilimab: 10mg/kg, administered D1, Q3W;
  * capecitabine: 1000 mg/m2 orally, D1-14, Q3W, twice daily;
  * bevacizumab injection: 7.5mg/kg, IV, D1, Q3W.
  Interventions: Drug: Cadonilimab (AK104) combined with chemotherapy and bevacizumab

INTERVENTIONS:
Drug: Cadonilimab (AK104) combined with chemotherapy and bevacizumab — Participants receive Cadonilimab PLUS chemotherapy and bevacizumab of each 21-day cycle.
  Treatment period (4-8 cycles)：
  * Cadonilimab: 10mg/kg, intravenous infusion, D1, Q3W;
  * CapeOx chemotherapy regimen Q3W+ bevacizumab, Q3W:
  oxaliplatin: 130 mg/m2 intravenous infusion, D1, Q3W; capecitabine: 850 mg/m2 orally, D1-14, Q3W, twice daily; bevacizumab injection: 7.5mg/kg, IV, D1, Q3W. Maintenance treatment period：
  * Cadonilimab: 10mg/kg, administered D1, Q3W;
  * capecitabine: 1000 mg/m2 orally, D1-14, Q3W, twice daily;
  * bevacizumab injection: 7.5mg/kg, IV, D1, Q3W.

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Cadonilimab (AK104) combined with chemotherapy and bevacizumab as first-line treatment for patients with RAS mutated or right sided-metastatic MSS colorectal cancer

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and voluntarily sign a written informed consent form, which must be signed before the designated research procedures required for the study are carried out.
2. Age at the time of signing the Informed Consent Form (ICF) is ≥ 18 years old and ≤ 75 years old, both male and female.
3. The Eastern Cancer Collaborative Organization (ECOG) has a physical fitness score of 0 or 1.
4. The expected survival period is ≥ 3 months.
5. Recurrent or incurable metastatic colorectal adenocarcinoma confirmed by Histopathology.(UICC/AJCC colorectal TNM stage System (8th edition 2017))
6. Genetic testing revealed RAS (including KRAS and NRAS) mutations, or primary sites located in the right half of the colon (including cecum, rising Colon and proximal 2/3 transverse colon).
7. Did not receive systemic treatment for recurrent or metastatic disease.
8. According to the RECIST v1.1 standard, there is at least one measurable tumor lesion. Agree to provide archived or freshly obtained tumor tissue samples (formalin fixed paraffin embedded [FFPE] tissue wax blocks or at least 5 unstained tumor tissue slice samples) to confirm PD-L1 expression.
9. The time interval between the end of adjuvant therapy was >12 months.
10. Having good organ function:

    1. Blood routine examination (no blood components or cell growth factors were used to support treatment within the first 7 days of randomization):

       * Absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L;
       * Platelet count ≥ 100 × 10^9/L;
       * Hemoglobin ≥ 9.0g/dL.
    2. Kidney:

       Creatinine<1.5 × ULN, or creatinine clearance rate * (CrCl) calculated value ≥ 50mL/min;

       *The Cockcroft Fault formula will be used to calculate CrCl: CrCL (mL/min)={(140 age) × Body weight (kg) × F} /(SCr (mg/dL) × 72) Among them: F=1 for males and F=0.85 for females; SCr=serum creatinine. Urinary protein<2+or 24-hour urine protein quantification<1.0g.
    3. Liver:

       Serum total bilirubin (TBiL) ≤ 1.5 × ULN; AST and ALT ≤ 2.5 × ULN (AST and ALT ≤ 5 for subjects with liver metastasis) × ULN, but not accompanied by elevated bilirubin);
    4. Coagulation function:

       International standardized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN
    5. Thyroid function: thyroid stimulating hormone (TSH) ≤ ULN; If abnormal, T3 and T4 levels should be investigated, and normal levels Can be selected
11. Female subjects with fertility must undergo a serum pregnancy test within 72 hours before the first medication, and the result should be negative. If a female subject with fertility engages in sexual activity with an unsterilized male partner, the subject must adopt an acceptable contraceptive method starting from screening and must agree to continue using the contraceptive method for 120 days after the last dose of the study drug; Periodic abstinence and safe period contraception are unacceptable contraceptive methods. Whether to stop contraception after this time point should be discussed with researchers.

    1. Women with fertility refer to those who have not undergone surgical sterilization (i.e. bilateral fallopian tube ligation, bilateral oophorectomy, or total hysterectomy) or those who have not undergone menopause (defined as those who have ceased menstruation for at least 12 consecutive months without alternative medical reasons, and whose serum follicle stimulating hormone levels are within the laboratory reference range of postmenopausal women);
    2. An efficient contraceptive method refers to a contraceptive method with a low failure rate (such as less than 1% per year) under continuous and correct use. Not all contraceptive methods are efficient. In addition to barrier contraception, female subjects with fertility can also use hormonal contraception (such as birth control pills), intrauterine device contraception, etc. to ensure that pregnancy does not occur.

Exclusion Criteria:

1. Previously received treatment with PD-1 monoclonal antibody, PD-L1 monoclonal antibody, or CTLA-4 monoclonal antibody.
2. The tumor tissue was found to be dMMR or MSI-H
3. Received palliative local treatment within the first 2 weeks of randomization; Received systemic non-specific immunomodulatory therapy (such as interleukin, interferon, thymosin, etc.) within the first 2 weeks of randomization; In the first 2 weeks of randomization, they received Chinese herbal medicine or traditional Chinese patent medicines and simple preparations with anti-tumor indications.
4. Currently participating in another clinical study, unless it is an observational, non-interventional clinical study, or a follow-up period of an intervention study.
5. Had or was currently present with other malignancies within the first 3 years of randomization. The following conditions can be included: cured uterus cervical carcinoma in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (cancer in situ) and T1 (tumor infiltrating basal membrane)].
6. Have active or untreated brain metastases, meningeal metastases, spinal cord compression, or leptomeningeal diseases. However, participants who meet the following requirements and have measurable lesions outside the central nervous system are allowed to be enrolled: asymptomatic after treatment, imageologically stable for at least 4 weeks before the start of study treatment (if there are no new or expanded brain metastases), and have stopped systemic glucocorticoid and anticonvulsant drug treatment for at least 2 weeks.
7. Have clinical symptoms of pleural effusion, pericardial effusion, or pleural/ascites that require frequent drainage (≥ once per month).
8. Active autoimmune diseases that require systematic treatment within the first 2 years of randomization, or autoimmune diseases that the researcher determines may recur or plan treatment. Except for the following:

   1. Skin diseases that do not require systematic treatment (such as vitiligo, alopecia, psoriasis, or eczema);
   2. Hypothyroidism caused by autoimmune thyroiditis requires only stable doses of hormone replacement therapy;
   3. Type I diabetes requiring only a stable dose of insulin replacement therapy;
   4. Childhood asthma has completely relieved, and no intervention is required in adulthood;
   5. Researchers have determined that the disease will not recur without external triggering factors.
9. Any of the following cardiovascular or cerebrovascular diseases or risk factors:

   1. Myocardial infarction, unstable angina, cerebrovascular accident, transient ischemic attack, acute or persistent myocardial ischemia, symptomatic heart failure (grade 2 or above according to the New York Heart Association functional classification), symptomatic or poorly controlled arrhythmia, or any arterial thromboembolism event occurred within the first 6 months of randomization.
   2. A history of deep vein thrombosis, pulmonary embolism, or other severe thromboembolism within the first 3 months of randomization.
   3. Have major vascular diseases such as aortic aneurysm, aortic dissection aneurysm, internal carotid artery stenosis that may endanger life or require surgery within 6 months.
   4. Uncontrolled hypertension (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg after standard antihypertensive therapy)
   5. Previous history of myocarditis and cardiomyopathy.
   6. Left ventricular ejection fraction (LVEF)<50%.
10. Toxicity that has not been alleviated by previous anti-tumor therapy is defined as failure to regress to the National Cancer Institute Adverse Event General Terminology Standard ((NCICTCAE v5.0) level 0 or 1, or the level specified in the inclusion/exclusion criteria, except for hair loss/pigmentation, ≥ Level 2 peripheral nerve disease).
11. The presence of interstitial lung disease or non infectious pneumonia is known, and the disease is currently symptomatic or requires systemic glucocorticoid treatment in the past. Researchers have determined that it may affect the toxicity assessment or management related to the study treatment.
12. Active pulmonary tuberculosis is known to exist. Subjects suspected of active pulmonary tuberculosis need to undergo chest X-ray examination, sputum examination, and elimination through clinical symptoms and signs.
13. Received systemic anti infective therapy (excluding antiviral therapy for hepatitis B or C) within the first 2 weeks of randomization.
14. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
15. Imaging (CT or MRI) shows that the tumor has invaded the large blood vessels or is not clearly delimited from the blood vessels.
16. Have clinical active diverticulitis, abdominal abscess, and gastrointestinal obstruction, unhealed wounds, ulcers, or fractures.
17. Clinically significant bleeding symptoms or bleeding tendencies within the first month of randomization, such as gastrointestinal bleeding, active hemoptysis, or bleeding, clotting disease are taking warfarin, aspirin, or other antiplatelet drugs (except maintenance doses: aspirin ≤100mg/ day, clopidogrel ≤75mg/ day), or regardless of severity，Subjects with any signs of bleeding or medical history that the investigator has determined are not suitable for enrollment.
18. Received major surgical treatment, open biopsy, or significant traumatic injury (except needle biopsy or gastroenteroscopic tissue biopsy) within the first 28 days of randomization.
19. Individuals with a known history of immune deficiency or HIV testing positive,Known active syphilis infection.
20. Subjects who require systemic treatment with glucocorticoids (>10mg/day prednisone or equivalent dose) or other immunosuppressive drugs within the first 14 days of randomization. Except for the following:

    1. If there is no active autoimmune disease, it is allowed to use inhaled, ophthalmic, or topical corticosteroids or other corticosteroids with a dose ≤ 10mg/day of prednisone or equivalent.
    2. The dosage of systemic glucocorticoids in physiological doses is ≤ 10mg/day of prednisone or equivalent doses of other glucocorticoids.
    3. Glucocorticoids are used as pretreatment for infusion related reactions or allergic reactions (such as medication before CT examination).
21. For untreated active hepatitis B subjects (HBsAg positive and HBV-DNA more than 1000 copies/ml [200IU/ml] or higher than the lower detection limit), patients with hepatitis B are required to receive anti hepatitis B virus treatment during the study treatment period; Active hepatitis C subjects (with positive HCV antibodies and HCV-RNA levels above the detection limit).
22. Received live vaccine within 30 days prior to randomization, or planned to receive live vaccine during the study period.
23. Subjects who have a known history of allergic or hypersensitive reactions to Cadonilimab, bevacizumab, capecitabine, oxaliplatin or any of their components. A history of severe hypersensitivity to other monoclonal antibodies is known.
24. In the judgment of the investigator, there is a concomitant disease that seriously endangers the safety of the subjects or interferes with the completion of the study, or subjects who were not suitable for inclusion for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Investigator | Up to approximately 1 year
  PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥ 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions was also considered PD. The PFS per RECIST 1.1 as assessed by Investigator will be presented.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) Per RECIST 1.1 as Assessed by Investigator | Up to approximately 1years
  ORR is defined as the percentage of the participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters).
Disease control Rate (DCR) Per RECIST 1.1 as Assessed by Investigator | Up to approximately 1 year
  DCR is the rate of CR,PR plus SD
Duration of Response (DoR) Per RECIST 1.1 as Assessed by Investigator | Up to approximately 1 year
  For participants who demonstrate CR or PR, DOR is defined as the time from first documented evidence of CR or PR until disease progression or death. The DOR per RECIST 1.1 as assessed by Investigator will be presented.
Time to response（TTR） | Up to approximately 6 months
  The time from randomization to the first CR or PR recorded
Overall Survival (OS) | From randomization through 90 days after last dose of study treatment
  OS is defined as the time from randomization to death due to any cause.
Number of Participants Who Experience an Adverse Event (AE) | From randomization through 30 days after last dose of study treatment
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be presented.
Number of Participants Who Experience a Serious AE (SAE) | From randomization through 90 days after last dose of study treatment
  An SAE is defined as any untoward medical occurrence that, at any dose: a.) Results in death; b.) Is life-threatening; c.) Requires inpatient hospitalization or prolongation of existing hospitalization; d.) Results in persistent or significant disability/incapacity; e.) Is a congenital anomaly/birth defect; f.) Other important medical events; h.) Is a new cancer (that is not a condition of the study) or i.) Is associated with an overdose. The number of participants who experience an SAE will be presented.

CONTACTS AND LOCATIONS:
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: Yes